CLINICAL TRIAL: NCT04697303
Title: Cross-sectional Study of Anorectal Function and Quality of Life in Patients With Middle and Low Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Quan Wang (Other)
Responsible Party: Sponsor-Investigator, Quan Wang, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: STARS-RC01
Record Dates: First submitted 2021-01-01; First posted 2021-01-06 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Middle and low rectal cancer
  Interventions: Other: anorectal function test

INTERVENTIONS:
Other: anorectal function test — anorectal function test

SUMMARY:
Understanding the quality of life and anorectal function changes in patients with middle and low rectal cancer after surgery can guide patients to recover after surgery and provide a valuable reference for surgeons in the selection of surgical methods. The purpose of this study is to: (1) Investigate the complication rate, recurrence and metastasis rate and survival of patients with middle and low rectal cancer. (2) QLQ-C30 and QLQ-CR29 questionnaires were used to assess the quality of life of patients with low- and middle-level rectal cancer at different periods after surgery. (3) Wexner constipation score and LARS syndrome score for anorectal function after operation for low rectal cancer. (4) The CIPE ejaculatory function score, IIEF-5 International Erectile Function Score, and FSFI-6 Female Sexual Function Index were used to assess the changes in sexual function of patients with low- and middle-position rectal cancer after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative patients with middle rectal cancer
2. Postoperative patients with low rectal cancer

Exclusion Criteria:

(1)Patients refused to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postoperative patients with middle and low rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | five years after the operation
  defined as time from the date of sugery to death

SECONDARY OUTCOMES:
QLQ-C30 | Every three months after the operation
  the score of Quality of life questionnaire QLQ-C30
QLQ-CR29 | Every three months after the operation
  the score of Quality of life questionnaire QLQ-C29
Wexner | Every three months after the operation
  the score of questionnaire Wexner
LARS | Every three months after the operation
  the score of questionnaire LARS
IIEF-5 | Every three months after the operation
  the score of questionnaire IIEF-5
CIPE | Every three months after the operation
  the score of questionnaire CIPE
FSFI-6 | Every three months after the operation
  the score of questionnaire FSFI-6

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin University First Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No